CLINICAL TRIAL: NCT03550716
Title: Surgical Sperm Retrieval in Non-obstructive Azoospermic Men: Microdissection Testicular Sperm Extraction vs. Multiple Needle-pass Percutaneous Testicular Sperm Aspiration
Brief Title: Surgical Sperm Retrieval in Non-obstructive Azoospermic Men: mTESE vs. TESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Holbaek Sygehus (Other); Skane University Hospital (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Christian Fuglesang S. Jensen, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-16033784
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Non-obstructive Azoospermia
Keywords: azoospermia; microdissection testicular sperm extraction; testicular sperm aspiration; male infertility; surgical sperm retrieval
MeSH Terms: conditions — Azoospermia; Infertility, Male

STUDY DESIGN:
Intervention Model Description: Trial type:
  Clinical randomized multi-center controlled trial
  Randomization:
  Block randomization is performed with the use of a computer generated block randomization list
  Participants:
  Patients with NOA undergoing fertility treatment
Who Masked: Participant
Masking Description: The randomization will be performed when the patient is asleep.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mTESE (Active Comparator): Patients randomized to mTESE
  Interventions: Procedure: mTESE
- TESA (Active Comparator): Patients randomized to TESA
  Interventions: Procedure: TESA

INTERVENTIONS:
Procedure: mTESE — mTESE is performed according to the initial description by Schlegel (4). General anesthesia is used. Midline incision of the scrotum is made and carried down to the level of the tunica vaginalis, which is opened to deliver the testis. Equatorial incision is made and the testis bivalved. The operating microscope is used to identify plump-appearing seminiferous tubules, and biopsies are taken from these areas. These samples are examined by an embryologist in the operating room after initial gross dispersion by passing the tissue through a 24G angiocatheter. The procedure is stopped if spermatozoa are found. If no plump tubules are found, random biopsies targeting every area of the testis are taken. If necessary the procedure is carried out on the contralateral testis. Hemostasis is obtained with careful bipolar cautery, and the tunica albuginea and the tunica vaginalis are closed with a running 4-0 Vicryl. Standard scrotal closure is performed and gentle pressure dressing is applied.
  Other Names: Microdissection testicular sperm extraction
  Arms: mTESE
Procedure: TESA — In general anesthesia an 18 gauge needle is introduced into each testis, and negative pressure applied with a 10 ml syringe. Multiple passes throughout the entire testis, numbering 50-100 passes, are made through a single percutaneous/tunical entry and continued until tissue is visible in the hub of the needle. This is removed by brisk extraction of the needle and pressure held to tamponade bleeding. The aspirated tissue is examined by an embryologist in the operating room after initial gross dispersion by passing the tissue through a 24 gauge angiocatheter.
  Other Names: Percutaneous testicular sperm aspiration
  Arms: TESA

SUMMARY:
Infertility is a significant social- and health problem in the Western World and at the moment in Denmark one in ten babies are born with the help of assisted reproduction. In 50% of infertile couples a male factor can be identified as a contributing cause (1).

Azoospermia is defined as the absence of spermatozoa in the ejaculate and it is a condition affecting 10-15% of infertile men (2, 3). Azoospermia is divided into obstructive azoospermia (OA) and nonobstructive azoospermia (NOA) of which the latter constitutes 60% (2, 3). In NOA the production of spermatozoa in the testis is either absent or markedly decreased.

Since 1999 microdissection testicular sperm extraction (mTESE) has become the preferred treatment option for NOA in many centers worldwide (4). The procedure is performed in general anesthesia using an operating microscope to carefully examine the entire testicular tissue for the presence of spermatozoa which can be used for assisted reproduction.

An alternative to mTESE is a percutaneous testicular sperm aspiration (TESA) or needle biopsy. This procedure is simple to perform using a biopsy needle to aspirate testicular tissue. The aspirated tissue is examined for the presence of spermatozoa that can be used in assisted reproduction.

Today there is no robust evidence on the optimal sperm retrieval protocol on men with NOA. This is in part due to the fact that no randomized trials have been performed to compare procedures. This study is the first to randomize procedures for surgical sperm retrieval.

Hypothesis In men with NOA, the investigators hypothesize that TESA is a viable first line approach compared to mTESE in regards to success rates of finding spermatozoa, complication rates and pregnancy outcomes.

A total of 110 men will be randomized to either mTESE or TESA and the rates of finding spermatozoa will be compared. However, for ethical reasons, because some believe mTESE have a greater chance of finding sperm cells, all men with a failed TESA will have a mTESE afterwards.

DETAILED DESCRIPTION:
Background Infertility is a significant social- and health problem in the Western World and at the moment in Denmark one in ten babies are born with the help of assisted reproduction. In 50% of infertile couples a male factor can be identified as a contributing cause (1).

Azoospermia is defined as the absence of spermatozoa in the ejaculate and it is a condition affecting 10-15% of infertile men (2, 3). Azoospermia is divided into obstructive azoospermia (OA) and nonobstructive azoospermia (NOA) of which the latter constitutes 60% (2, 3). In NOA the production of spermatozoa in the testis is either absent or markedly decreased.

Since 1999 microdissection testicular sperm extraction (mTESE) has become the preferred treatment option for NOA in many centers worldwide (4). The procedure is performed in general anesthesia using an operating microscope to carefully examine the entire testicular tissue for the presence of spermatozoa which can be used for intracytoplasmic sperm injection (ICSI). The advantages of mTESE include high sperm retrieval rates (SRR), in recent systematic reviews reported around 52% (5-8), and low reported complication rates (9-11). However mTESE is a time-consuming invasive procedure requiring the right expertise, the right equipment and a proper setup of the fertility clinic.

An alternative to mTESE is a percutaneous testicular sperm aspiration (TESA). This procedure is simple to perform using a biopsy needle to aspirate testicular tissue. The aspirated tissue is examined for the presence of spermatozoa and SRR for this procedure is usually reported around 25% (5-8). The lower SRR compared to mTESE is the main limitation of this method, but the procedure is well tolerated by patients and due to its simplicity and short duration it can easily be performed in the out-patient clinic. In collaboration with University of Michigan the TESA technique has been improved by using an 18 gauge needle and performing multiple (50-100) passes throughout the entire testicular tissue while applying a vacuum. In the remainder of this document this multiple needle-pass TESA will be referred to as "TESA". Recently the investigators retrospectively evaluated this approach and found a SRR of 30% using TESA and interestingly the SRR of mTESE following a failed TESA was only 11% (12).

However, there is no robust evidence on the optimal sperm retrieval protocol on men with NOA. This is in part due to the fact that no randomized trials have been performed to compare the two procedures. Often patients from different countries are required to pay the infertility treatment themselves and the cost for a TESA is around $500 while a mTESE is around $8.000. This makes it difficult to perform a randomized trial in most countries but because of the public health systems of Denmark and Sweden there is a unique possibility to be the first in the world to do a randomized trial on this matter.

Hypothesis In men with NOA, the investigators hypothesize that TESA is a viable first line approach compared to mTESE in regards to SRR, complication rates and pregnancy outcomes.

Screening and randomization Potential study patients and their partners will initially be identified in their work-up during their infertility treatment. When a patient is identified as having NOA, the patient will be screened according to inclusion- and exclusion criteria. If these are met and the patient provides an informed consent for participation, the patient is included and randomized to undergo mTESE or TESA. Patients will be recruited from the fertility clinics at Herlev and Gentofte Hospital, Malmö University Hospital, Holbaek Hospital and Rigshospitalet in collaboration with Department of Growth and Reproduction, Rigshospitalet.

Planning the treatment and surgery Treatment of the infertile couples will follow regular treatment protocols at the respective fertility clinics. This includes freezing retrieved sperm cells and thawing them in relation to the oocyte retrieval. As an alternative to sperm cell freezing, retrieved oocytes will be frozen and thawed in relation to the surgical sperm retrieval. The aim is to have 6-8 oocytes stored before operation for couples following this route. All patients will undergo full anesthesia. If the patient is randomized to TESA and this fails, then a salvage mTESE can be done immediately while in the operating theatre.

Visits Before visit 1 all patients and their partners will have received written and oral information on the study and will have had time to provide an informed consent.

At visit 1 patients and possibly their partners (mandatory in cases of oocyte cryopreservation) meet with the primary investigator. It will be secured that an informed consent for participation is signed. The focus of visit 1 will be on accessing the men's evaluation leading to the NOA diagnosis and checking inclusion- and exclusion criteria. In addition, information regarding medical history will be obtained and a physical examination of the external genitalia will be carried out. Patients will fill out questionnaires on psychosexual health and pain before the visit and their answers will be reviewed together. A blood sample will be taken for the purpose of measuring hormone levels and for storage in the biobank. Likewise patients will bring a semen sample for storage in the biobank. If not previously done patients will be tested with regards to karyotype, AzF microdeletions and CFTR mutations if deemed necessary.

Visit 2 will be the actual procedure. Follow-up is comprised by patients filling out the mentioned questionnaires, reporting any complications and having a blood sample drawn at visit 3 and 4. Follow-up will primarily be done by phone/mail, but at visit 3 and 4 patients will have to go to the Department of Growth and Reproduction, Rigshospitalet (for Danish patients) or the fertility clinic at Malmö University Hospital (for Swedish patients) to have blood samples drawn. Samples collected in Sweden will be send for analysis at the Department of Growth and Reproduction, Rigshospitalet. Pregnancy outcome will be reported by phone/mail 9-15 months after the procedure is done.

Biobank A research biobank will be made containing blood samples, semen and testicular tissue. Blood samples will be used for genotyping and to measure relevant biomarkers including piRNAs, miRNAs, protein markers and biochemical markers. Semen will also be used to measure relevant biomarkers. Testicular tissue will be used for testing for molecular and biochemical markers of spermatogenesis and to measure intratesticular testosterone levels. Additionally testicular tissue showing maturation arrest will be used for attempts to maturate germ cells in vitro (not to be used for fertilization, only research). The purpose of the above is to find markers of successful sperm retrieval and to get a better understanding of the biology of NOA and potentially to develop pharmacological strategies in the future for treating certain forms of NOA as e.g. maturations arrest.

Safety and adverse events:

Hematoma As TESA/ mTESE is a surgery there is a risk of post-operative bleeding leading to scrotal or spermatic cord hematomas. Estimated risk <1,5%.

Infection As TESA/ mTESE is a surgery there is a risk of infection. Estimated risk <1% Pain Pain is expected to occur after both procedures but especially after mTESE Drop in testosterone level In the litterature this is reported as a transient event following mTESE however there is a risk of more lasting androgen deficiency. Careful surgical techniques will be used to limit the amount of tissue damage.

Possible disadvantages:

Lower SRR following TESA SRR are reported lower for TESA compared to mTESE. For this reason patients with an unsuccessful TESA will be offered a salvage mTESE Oocyte cryopreservation In the past fertilization outcomes after cryopreservation have been lower compared to fresh oocytes. However with the evolution of cryopreservation techniques (vitrification) IVF pregnancy rates with the use of cryopreserved oocytes are now similar to those of fresh oocytes. (15) Grading of complications Complications will be graded according to the Clavien-Dindo classification of surgical complications (14).

Ethical evaluation This study will follow the newest edition of the Helsinki Declaration and at all times follow applicable laws. It will be reported to "Datatilsynet", "Videnskabsetisk komite" and the "Ethical Committee of Lund University".

Some of the ethical aspects related to this project have been briefly described in the safety and adverse events section. Both mTESE and TESA are safe procedures and although the investigators previously found a higher complication rate with mTESE compared to TESA (12), the general literature describe both procedures with comparable risks related to infection and hematomas.

To make the study possible to complete, either the sperm cells or the oocytes retrieved from the women will have to undergo cryopreservation. Sperm cell cryopreservation is standard practice at the fertility clinics today. Previously only fresh oocytes were used for in-vitro fertilization but recently it has been shown that treatment using cryopreserved oocytes give similar pregnancy rates to those of fresh oocytes. Thus freezing the oocytes should not be a disadvantage to the couples.

When looking at sperm retrieval rates, mTESE has until now been superior to TESA. However with the improved TESA results are expected to be more equal. In addition patients randomized to TESA will have the benefit of a more simple and less invasive treatment compared to mTESE. Moreover patients randomized to TESA will be provided with an option to receive a salvage mTESE that can be carried out the same day because all patients will undergo full anesthesia. In this way all patients included in the study will receive equal treatment options for NOA.

Attempts of maturation of germ cells in vitro will be made using tissue with partial or total maturation arrest. If successful, the germ cells maturated in vitro will not be used for any attempt of fertilization but only as "proof of concept" regarding treatment of azoospermia due to maturation arrest.

In a broader picture this project will be the first randomized study on this matter and therefore it will bring a clearer picture on which is the optimal sperm retrieval technique for men with NOA. This will benefit many patients with NOA in the future.

Publication of results:

Results from the study will be published in international peer-reviewed scientific journals, national journals and hospital websites. This will happen no matter the outcome of the study meaning that both positive, negative and inconclusive results will be made public. Additionally results will be presented at conferences and meetings. All published results will be made anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Azoospermia verified in at least two semen samples within the past six months, including assessment of the centrifuged pellet as per the WHO 5th edition (13)
* Testis volume (Prader's orchidometer) ≤ 15ml on both sides
* No indication of obstructive causes of azoospermia in medical history or physical examination (ex. absent vas deferens, vasectomy, scrotal trauma/injury, hernia repair or other operations potentially damaging the vas deferens)
* Capable and legally competent individual

Exclusion Criteria:

* Previous attempts of surgical sperm retrieval
* Previous testicular biopsy
* Anejaculation
* Retrograde ejaculation
* Bleeding disorders rendering surgery too high a risk
* Klinefelters Syndrome
* XX male
* AZFa/b microdeletion
* CFTR mutation
* Inability to understand and/or stick to the written information
* Patients not deemed suitable for general anesthesia

Exclusion during follow-up

* A patient can at any time during the study withdraw their consent of participation
* Normal histology on testis biopsy following TESA or mTESE

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 46XY
Enrollment: 110 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval rate | Assessed immediately after the procedure
  Rate of succesful sperm retrievals defined as at least one spermatozoa found suitable for intracytoplasmic sperm injection (ICSI)

SECONDARY OUTCOMES:
Conversion rate to mTESE | Recorded immediately after the procedure
  Rate of conversion from TESA to mTESE in the TESA group
Sperm retrieval rate after salvage mTESE | Recorded immediately after the procedure
  Rate of succesful sperm retrievals following salvage mTESE
Complication rates | Recorded in the first 6 months after surgery
  Any complication after surgery
Pregnancy outcomes | Recorded in the first 9-15 months after surgery
  Fertilization rate (per injected oocyte), chemical pregnancy rate, clinical pregnancy rate and live birth rate (per IVF cycle)
Difference in perceived stress scale (PSS) score | Three months before to three months after surgery
  The validated questionnaire PSS measures the perception of stress. The scale range is 0-40 with a higher score indicating more perceived stress.
Difference in PainDetect pain scale score | Three months before to three months after surgery
  Based on the validated questionnaire PainDetect. The scale range is 0-38 with a higher score indicating a larger neuropathic pain component
Difference in pain score - Visual Analog Scale | Three months before to three months after surgery
  Pain reported on the visual analog scale with the range 0-10. A higher score indicates more pain.
Difference in erectile function score | Three months before to three months after surgery
  Based on the validated questionnaire the International Index of Erectile Function (IIEF-5). The scale range is 5-25 with a higher score indicating a better erectile function.
Difference in Hospital Anxiety and Depression Scale (HADS) scores - subscale anxiety. | Three months before to three months after surgery
  Anxiety measured with the validated questionnaire HADS. The subscale range is 0-21 with a higher score indicating more anxiety.
Difference in Hospital Anxiety and Depression Scale (HADS) scores - subscale depression. | Three months before to three months after surgery
  Depression measured with the validated questionnaire HADS. The subscale range is 0-21 with a higher score indicating more depresssion.
Difference in Short-Form 12-item Survery (SF-12) mental health summary score | Three months before to three months after surgery
  Mental Health Composite Scores (MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Difference in Short-Form 12-item Survery (SF-12) physical health summary score | Three months before to three months after surgery
  Physical Health Composite Scores (PCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of Health measured by the scales and 100 indicates the highest level of health.
Age as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Age
Body Mass Index (BMI) as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  BMI
Testis histology as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Testis Histology
Testis size as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Testis size
Biomarkers as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Relevant (not identified yet) biomarkers in blood, seminal fluid and/or testicular tissue,
Intra-testicular testosterone level as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Intra-testicular testosterone level
FSH as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Follicle-stimulating hormone level
LH as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Luteinizing hormone level
Testosterone as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Testosterone level
Inhibin B as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Inhibin B level
AMH as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Anti-Müllerian hormone level
Estradiol as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Estradiol level
Prolactin as a predictor of successful sperm retrieval | Calculated 1-3 years after surgical intervention
  Baseline Prolactin level

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Holbæk Sygehus, Holbæk
- Malmö University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharlip ID, Jarow JP, Belker AM, Lipshultz LI, Sigman M, Thomas AJ, Schlegel PN, Howards SS, Nehra A, Damewood MD, Overstreet JW, Sadovsky R. Best practice policies for male infertility. Fertil Steril. 2002 May;77(5):873-82. doi: 10.1016/s0015-0282(02)03105-9. No abstract available. PMID 12009338
- [Background] Jarow JP, Espeland MA, Lipshultz LI. Evaluation of the azoospermic patient. J Urol. 1989 Jul;142(1):62-5. doi: 10.1016/s0022-5347(17)38662-7. PMID 2499695
- [Background] Willott GM. Frequency of azoospermia. Forensic Sci Int. 1982 Jul-Aug;20(1):9-10. doi: 10.1016/0379-0738(82)90099-8. No abstract available. PMID 7095683
- [Background] Schlegel PN. Testicular sperm extraction: microdissection improves sperm yield with minimal tissue excision. Hum Reprod. 1999 Jan;14(1):131-5. doi: 10.1093/humrep/14.1.131. PMID 10374109
- [Background] Dabaja AA, Schlegel PN. Microdissection testicular sperm extraction: an update. Asian J Androl. 2013 Jan;15(1):35-9. doi: 10.1038/aja.2012.141. Epub 2012 Dec 17. PMID 23241638
- [Background] Deruyver Y, Vanderschueren D, Van der Aa F. Outcome of microdissection TESE compared with conventional TESE in non-obstructive azoospermia: a systematic review. Andrology. 2014 Jan;2(1):20-4. doi: 10.1111/j.2047-2927.2013.00148.x. Epub 2013 Nov 6. PMID 24193894
- [Background] Donoso P, Tournaye H, Devroey P. Which is the best sperm retrieval technique for non-obstructive azoospermia? A systematic review. Hum Reprod Update. 2007 Nov-Dec;13(6):539-49. doi: 10.1093/humupd/dmm029. Epub 2007 Sep 24. PMID 17895238
- [Background] Bernie AM, Mata DA, Ramasamy R, Schlegel PN. Comparison of microdissection testicular sperm extraction, conventional testicular sperm extraction, and testicular sperm aspiration for nonobstructive azoospermia: a systematic review and meta-analysis. Fertil Steril. 2015 Nov;104(5):1099-103.e1-3. doi: 10.1016/j.fertnstert.2015.07.1136. Epub 2015 Aug 8. PMID 26263080
- [Background] Amer M, Ateyah A, Hany R, Zohdy W. Prospective comparative study between microsurgical and conventional testicular sperm extraction in non-obstructive azoospermia: follow-up by serial ultrasound examinations. Hum Reprod. 2000 Mar;15(3):653-6. doi: 10.1093/humrep/15.3.653. PMID 10686214
- [Background] Okada H, Dobashi M, Yamazaki T, Hara I, Fujisawa M, Arakawa S, Kamidono S. Conventional versus microdissection testicular sperm extraction for nonobstructive azoospermia. J Urol. 2002 Sep;168(3):1063-7. doi: 10.1016/S0022-5347(05)64575-2. PMID 12187223
- [Background] Ramasamy R, Yagan N, Schlegel PN. Structural and functional changes to the testis after conventional versus microdissection testicular sperm extraction. Urology. 2005 Jun;65(6):1190-4. doi: 10.1016/j.urology.2004.12.059. PMID 15922422
- [Background] Jensen CF, Ohl DA, Hiner MR, Fode M, Shah T, Smith GD, Sonksen J. Multiple needle-pass percutaneous testicular sperm aspiration as first-line treatment in azoospermic men. Andrology. 2016 Mar;4(2):257-62. doi: 10.1111/andr.12143. Epub 2016 Jan 20. PMID 26789006
- [Background] WHO laboratory manual for the examination and processing of human semen. World Health Organization. 2010;5th ed.
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Argyle CE, Harper JC, Davies MC. Oocyte cryopreservation: where are we now? Hum Reprod Update. 2016 Jun;22(4):440-9. doi: 10.1093/humupd/dmw007. Epub 2016 Mar 22. PMID 27006004